CLINICAL TRIAL: NCT01080924
Title: Demonstration of Broncholytic Effects in Subjects With Obstructive Airway Diseases by Low Frequency Ultrasound
Acronym: Pabes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fraunhofer-Institute of Toxicology and Experimental Medicine (Other)
Collaborators: Institute for Pharmacology and Toxicology, RWTH Aachen (Unknown)
Responsible Party: Prof. Dr. Jens Hohlfeld, Fraunhofer-Institute of Toxicology and Experimental Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 08/10 Pabes
Record Dates: First submitted 2010-03-03; First posted 2010-03-05 (Estimated); Last update posted 2011-06-27 (Estimated); Status verified 2011-06

CONDITIONS: Healthy Volunteers; COPD GOLD I to IV; Asthma GINA 1 to 4

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Low frequency ultrasound spectroscopy (Experimental): Low frequency ultrasound spectroscopy after broncholysis
  Interventions: Device: Low frequency ultrasound spectroscopy after broncholysis

INTERVENTIONS:
Device: Low frequency ultrasound spectroscopy after broncholysis — Low frequency ultrasound spectroscopy is a novel non-invasive approach to real-time diagnostics of the lungs. Low frequency ultrasound at 10 to 1000 kHz permits monitoring of the air and water contents of the human thorax.

SUMMARY:
This study is aiming at evaluating whether low frequency ultrasound spectroscopy is a sensitive tool to detect broncholytic effects in patients with obstructive airway diseases.

ELIGIBILITY:
Inclusion Criteria:

* • 18 - 70 years

  * for the healthy cohort:

    * FEV1 > 80 % pred, FEV1/FVC ≥ 70 % pred., no history of allergies or asthma
    * nonsmokers, with a history of less than 1 packyear having been nonsmokers for at least the last five years
  * for the COPD cohort: COPD GOLD I to IV according to current guidelines (2)
  * for the asthma cohort: history of asthma GINA I to IV according to current guidelines (3)
  * BMI ≤ 30 kg/m2
  * Able and willing to give written informed consent
  * Available to complete all study measurements

Exclusion Criteria:

* • medical conditions which prohibit the use of salbutamol

  * recent exacerbation of COPD or asthma or lower respiratory tract infection (four weeks previous to informed consent visit)
  * past or present disease, which as judged by the investigator, may affect the outcome of the study. These diseases include, but are not limited to, cardiovascular disease, malignancy, hepatic disease, renal disease, hematological disease, neurological disease, psychiatric disease, endocrine disease or pulmonary disease (including but not confined to asthma, tuberculosis, bronchiectasis or cystic fibrosis)
  * history of drug or alcohol abuse which would interfere with the subject's proper completion of the protocol assignment
  * risk of non-compliance with study procedures
  * suspected inability to understand the protocol requirements, instructions and study-related restrictions, the nature, scope, and possible consequences of the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2010-02; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
• change of the difference of expiratory and inspiratory TOF Expectation: The difference of ex and inspiratory TOF should increase after broncholysis. A change above 10us will be considered significant | 10 minutes post broncholysis

CONTACTS AND LOCATIONS:
Overall Officials: Jens Hohlfeld, Prof. Dr., Principal Investigator — Fraunhofer Institute for Toxicology and Experimental Medicine
Locations (1):
- Fraunhofer ITEM, Hanover, Lower Saxony, Germany

REFERENCES:
- [Derived] Morenz K, Biller H, Wolfram F, Leonhadt S, Ruter D, Glaab T, Uhlig S, Hohlfeld JM. Detection of air trapping in chronic obstructive pulmonary disease by low frequency ultrasound. BMC Pulm Med. 2012 Mar 16;12:8. doi: 10.1186/1471-2466-12-8. PMID 22424178